CLINICAL TRIAL: NCT04826731
Title: Effect of Respiratory Exerciser on Pulmonary Functions of COVID-19 Patients, A Prospective Observational Study
Brief Title: Effect of Respiratory Exerciser on Pulmonary Functions of COVID-19 Patients
Status: Completed | Type: Observational
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Kerem Ensarioğlu, Medical Doctor, Diskapi Yildirim Beyazit Education and Research Hospital
Other Study IDs: 104/18
Record Dates: First submitted 2021-03-27; First posted 2021-04-01 (Actual); Results first posted 2022-01-31 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Covid19; Respiratory Function Loss; Coronavirus Infection; Pneumonia, Viral
Keywords: Pulmonary Rehabilitation; Respiratory Function Loss
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Pneumonia, Viral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Incentive Spirometer Group: Patients who would use an incentive spirometer, in addition to standard care provided to COVID-19 patients, will be categorized under "Incentive Spirometer Group".
  Interventions: Other: Incentive Spirometer/Respiratory Exerciser
- Standard Care Group: Patients who did not use an incentive spirometer despite being suggested to do so will be categorized under "Standard Care Group".

INTERVENTIONS:
Other: Incentive Spirometer/Respiratory Exerciser — A patient is considered acceptable for the "Incentive Spirometer Group" if the patient can use an incentive spirometer and/or a respiratory exerciser at least four times per day. A pulmonary medicine specialist will confirm the proper usage of the device.
  Groups: Incentive Spirometer Group

SUMMARY:
COVID-19 infection is the cause of the current pandemic, responsible for loss of life and disability at a rate unseen before. Among survivors, the infection may cause lasting damage, such as permanent loss of lung function.

This study aims to investigate if pulmonary rehabilitation done via supportive devices may reduce or prevent lung function injury. Patients will be chosen among COVID-19 patients who require hospitalization. Patients then will be divided into two groups, those who had used said devices, and compare them to those who had not used them for any reason. After a month, two groups will be evaluated by respiratory function tests, which are expected to provide the results required for a proper comparison.

Pulmonary rehabilitation provided by the supportive devices is expected to either lessen or eliminate a loss of pulmonary function over time, compared to the group who did not use them.

DETAILED DESCRIPTION:
SARS-CoV-2 is a novel coronavirus that is responsible for the current pandemic. Its clinical presentation varies from asymptomatic infection to severe respiratory failure requiring intensive care stay. Loss of respiratory function had been observed in survivors of other coronaviruses in earlier studies. The degree of respiratory function loss and if any intervention may reduce or prevent it remains an issue to be clarified.

The study's goal is to investigate the effects of pulmonary rehabilitation via a supporting device on COVID-19 patients during a follow-up period of one month. The primary method of investigation of pulmonary functions is comparing peak expiratory flow (PEF) at the time of diagnosis and after treatment.

The study hypothesizes that patients who had successfully used a respiratory exerciser or a similar aid device will have better PEF results at the end of the first-month evaluation.

The effect of an incentive spirometer and/or a respiratory exerciser on the pulmonary function results is the main element under investigation in this study. The hospital provides these devices, and in cases, patients demand another device, the patients and their relatives are asked to purchase such equipment.

Pulmonary function tests (PFT) are considered a part of routine evaluation for the COVID-19 patients a month after the treatment. Patients are considered suitable for PFT evaluation if the COVID-19 infectious process is deemed treated, and other contraindications for PFT are not present, such as recent surgery or pneumothorax.

Patients admitted to the pulmonary medicine ward for COVID-19 infection are generally those who already have respiratory comorbidity, including chronic obstructive pulmonary disease, asthma, concurrent pneumonia, and respiratory failure. Due to these reasons, PFT is not considered an acceptable evaluation method during the acute phase and is not requested. PEF testing, on the other hand, remains a simple yet effective alternative compared to PFT due to being more portable, the presence of disposable parts, and overall cost. It is the initial choice of evaluation for patients after a clinical response is seen to treatment and testing is deemed safe.

The respiratory exercise is considered a part of COVID-19 care, primarily due to patients' comorbidities, as mentioned above. This approach is limited in terms of healthcare personnel for on-point pulmonary rehabilitation due to both the disease's infectious nature and limited resources. Respiratory exercise devices are accepted as a reasonable alternative that can be quantitively monitored and provided on a daily basis.

This prospective study plans to evaluate the impact of respiratory exercise provided by incentive spirometers and respiratory exercisers. The evaluation will be performed by comparing the initial PEF result after the end of COVID-19 treatment and subsequent ward discharge; to the PEF result of the PFT evaluation at the end of the first month.

ELIGIBILITY:
Inclusion Criteria:

1. Being at least 18 years or older
2. Approval given both written and orally to the study participation
3. COVID-19 positivity proven by reverse transcription-polymerase chain reaction (RT-PCR) testing
4. At least one evaluation/consultation performed by a pulmonary medicine specialist OR admission to pulmonary medicine ward from another department in the hospital
5. First hospital admission has to be via emergency ward, regardless of the concurrent hospital stay.
6. Cooperation at an acceptable degree for pulmonary function testing.

Exclusion Criteria:

1. Any contraindication presence for pulmonary function testing (such as anatomic abnormalities, recent cardiac history, and severe respiratory failure)
2. Former COVID-19 history.
3. Persistent pulmonary or other systemic pathology (which prevents hospital discharge)
4. Refusal to participate in the monthly evaluation.
5. Persistent COVID-19 RT-PCR presence (which prevents PFT testing)
6. Known severe limitation in former PFT testing (FEV1 being lower than 30%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected among those who apply to emergency service and evaluated by a pulmonary medicine resident or specialist. Among this population, further selection will be performed via the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bahar Kurt, Professor, Principal Investigator — Dışkapı Yıldırım Beyazıt Training and Research Hospital Pulmonary Medicine
Locations (1):
- Dışkapı Yıldırım Beyazıt Training and Research Hospital Pulmonary Medicine Clinic, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be shared with other researchers working on a similar process, with proper credentials and acknowledgments given according to ICJME clinical trial registration policy. Signed Informed Consent Forms will only be shared with proper legal bodies and ethical committees in case of an ethical dilemma.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be available for the 6 months after initial publication.
Access Criteria: The information mentioned above will be shared upon contact with the corresponding author. The criteria for data sharing would be that the researchers making the request would preferably seek a similar goal in the study proposal.

REFERENCES:
- [Background] Torres-Castro R, Vasconcello-Castillo L, Alsina-Restoy X, Solis-Navarro L, Burgos F, Puppo H, Vilaro J. Respiratory function in patients post-infection by COVID-19: a systematic review and meta-analysis. Pulmonology. 2021 Jul-Aug;27(4):328-337. doi: 10.1016/j.pulmoe.2020.10.013. Epub 2020 Nov 25. PMID 33262076
- [Background] Gemicioglu B, Borekci S, Dilektasli AG, Ulubay G, Azap O, Saryal S. Turkish Thoracic Society Experts Consensus Report: Recommendations for Pulmonary Function Tests During and After COVID 19 Pandemic. Turk Thorac J. 2020 May;21(3):193-200. doi: 10.5152/TurkThoracJ.2020.20107. PMID 32584237
- [Background] Mo X, Jian W, Su Z, Chen M, Peng H, Peng P, Lei C, Chen R, Zhong N, Li S. Abnormal pulmonary function in COVID-19 patients at time of hospital discharge. Eur Respir J. 2020 Jun 18;55(6):2001217. doi: 10.1183/13993003.01217-2020. Print 2020 Jun. PMID 32381497
- [Background] Anastasio F, Barbuto S, Scarnecchia E, Cosma P, Fugagnoli A, Rossi G, Parravicini M, Parravicini P. Medium-term impact of COVID-19 on pulmonary function, functional capacity and quality of life. Eur Respir J. 2021 Sep 16;58(3):2004015. doi: 10.1183/13993003.04015-2020. Print 2021 Sep. PMID 33574080

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Incentive Spirometer Group | Standard Care Group
Started | 10 | 4
Completed | 10 (All patients were initially accepted as the study group per study design, with those unable to utilize respiratory exerciser (n=4) were later removed to standard care group.) | 4 (Patients who could not use the respiratory exerciser (n=2) or refused to do so (n=2) were accepted as the control group.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Initially, all fourteen patients were accepted as the study group, afterwards, those who had refused to or could not cooperate with the respiratory exerciser were accepted as the standard care group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Incentive Spirometer Group | Standard Care Group | Total
Number analyzed (Participants) | 10 | 4 | 14
Age, Continuous [Median (Full Range); unit: Years] | 54 [39 to 71] | 41 [39 to 75] | 51 [39 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 7 | 2 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Turkey | 10 | 4 | 14
Charlson Comorbidity Index [Median (Full Range); unit: Units on a scale] — Charlson Comorbidity Index is utilized for the evaluation of the total severity of comorbidities present on a patient. It calculates an estimated ten years survival rate, based on a point scale, with higher scores having increased overall mortality. The scale ranges beings from 0 points (98% ten years survival ) with 7 points presented with 0% 10 years survival, with the theoretical upper limit being 31 points (accumulation of all possible comorbidities). For this study's interest, 1 point presents with 96%, 2 with 90%, 3 with 77%, and 4 with 55% survival rate (highest score observed here)
  Units on a scale | 1 [0 to 3] | 0 [0 to 4] | 1 [0 to 4]
Peak Expiratory Flow (Hospital Discharge) [Median (Full Range); unit: ml/min] — Peak Expiratory Flow (PEF) is calculated by personal handheld devices given to the patients. The initial testing was performed at the time of hospital discharge, for which afterward respiratory exerciser was requested of the patients. This initial PEF value is accepted as the baseline measure for which the comparison was made at the follow-up (which was defined as the first evaluation performed one month after hospital discharge). The normal PEF range in ml/min depends on the patient's age and gender, with an estimated average of 571 ml/min in a 20-year-old, 175 cm male.
  ml/min | 80 [59 to 127] | 100 [45 to 105] | 86 [45 to 127]
Initial Oxygenation Requirement [Count of Participants; unit: Participants] — The initial oxygen requirement is defined as the oxygenation required for a patient to be considered stable (a saturation % of 90 or above) at the time of the first day of hospital admission. The categorization is made according to the delivery methods, with each method providing a certain oxygen flow. Nasal support includes 0-4 liter/min, mask category includes a support level of 4-10 l/min, and high flow definition supports any l/min above 10 l/min. Due to the study design of respiratory testing being performed at hospital discharge, these parameters were accepted as baseline results.
  Participants
    None | 4 | 1 | 5
    Nasal | 4 | 2 | 6
    Mask | 2 | 1 | 3
Maximum Oxygenation Requirement [Count of Participants; unit: Participants] — The maximum oxygenation requirement is defined as the highest oxygenation required for a patient to be considered stable (a saturation % of 90 or above). The categorization is made according to the delivery methods, with each method providing a certain oxygen flow. Nasal support includes 0-4 liter/min, mask category includes a support level of 4-10 l/min, and high flow definition supports any l/min above 10 l/min. Due to the study design of respiratory testing being performed at hospital discharge, these parameters were accepted as baseline results.
  Participants
    None | 0 | 1 | 1
    Nasal | 6 | 2 | 8
    Mask | 3 | 1 | 4
    High Flow | 1 | 0 | 1
Discharge Oxygenation Requirement [Count of Participants; unit: Participants] — The discharge oxygen requirement is defined as the oxygenation required for a patient to be considered stable (a saturation % of 90 or above) at the time of hospital discharge. The categorization is made according to the delivery methods, with each method providing a certain oxygen flow. Nasal support includes 0-4 liter/min, mask category includes a support level of 4-10 l/min, and high flow definition supports any l/min above 10 l/min. Due to the study design of respiratory testing being performed at hospital discharge, these parameters were accepted as baseline results.
  Participants
    None | 8 | 4 | 12
    Nasal | 2 | 0 | 2
    Mask | 0 | 0 | 0
Hospitalization Duration (Days) [Median (Full Range); unit: Days] — The hospitalization duration is accepted as a baseline parameter, as the respiratory exercise component of the study would begin at the time of patient discharge.
  Days | 10 [5 to 18] | 5 [3 to 13] | 8 [3 to 18]
Discharge to Follow-up Duration (Days) [Median (Full Range); unit: Days] | 31 [13 to 41] | 30 [29 to 35] | 30 [13 to 41]

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Expiratory Flow (Absolute Value)
Description: Two PEF results will be compared in the study. The first PEF testing will be performed by a handheld device and the second measurement will be performed either by an office spirometer or a handheld device. The priority will be given to the office spirometer for testing preference.
Time Frame: The first PEF testing will be performed seven days after initial diagnosis. The second testing will be performed one month after the hospital discharge, among those who are considered suitable for testing.
Population: Initially, all fourteen patients were accepted as the study group, among those four patients who could not utilize the respiratory exerciser device were later moved to the standard care group.
Measure: Median (Full Range); unit: ml/min
Arm/Group | Incentive Spirometer Group | Standard Care Group
Number analyzed (Participants) | 10 | 4
ml/min | 175 [40 to 320] | 160 [10 to 430]
Statistical Analysis 1: Comparison: Incentive Spirometer Group vs Standard Care Group; Nonparametric testing was utilized due to non-standard distribution and reduced sample size. Comparison between groups was made by Mann-Whitney U testing. Spearman's rho was utilized for correlation analysis. No subgroup analyses were planned for the study; Test type: Other; p = 0.374, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Change in Peak Expiratory Flow (Percentage)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Percentage of Predicted Value
Arm/Group | Incentive Spirometer Group | Standard Care Group
Number analyzed (Participants) | 10 | 4
Percentage of Predicted Value | 70 [27 to 178] | 51 [4 to 239]
Statistical Analysis 1: Comparison: Incentive Spirometer Group vs Standard Care Group; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.635, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Peak Expiratory Flow (Follow-up)
Description: The Peak Expiratory Flow (PEF) results were obtained at the follow-up evaluation. These results were then compared with the initial baseline measurement of PEF performed at the hospital discharge.
Time Frame: Testing for PEF results were performed at the follow-up evaluation, which was done 1 month post-baseline.
Population: as for baseline characteristics
Measure: Median (Full Range); unit: ml/min
Arm/Group | Incentive Spirometer Group | Standard Care Group
Number analyzed (Participants) | 10 | 4
ml/min | 400 [190 to 540] | 500 [260 to 610]

4. Secondary Outcome: Forced Expiratory Volume (FEV1)
Description: Forced Expiratory Volume (FEV1) result of the pulmonary function testing was to be used as a pulmonary function parameter. It was performed via standard office spirometry. It was calculated as an absolute value (in liters) and as a percentage (compared to the normal population data) It was to be used as a validation method to ensure patients did not have a former yet undiagnosed respiratory disease and to validate the presence of abnormal Peak Expiratory Flow (PEF) values.
Time Frame: Forced Expiratory Volume (FEV1) was evaluated at the follow-up evaluation, which was performed one-month post-baseline.
Population: Due to cooperation difficulties and/or differences above 10% in repeated testing, a total of 6 patients were excluded from the FEV1 evaluation.
Measure: Median (Full Range); unit: Percentage of Predicted Value
Arm/Group | Incentive Spirometer Group | Standard Care Group
Number analyzed (Participants) | 7 | 3
Percentage of Predicted Value | 70 [59 to 127] | 100 [60 to 105]

5. Secondary Outcome: Forced Vital Capacity (FVC)
Description: Forced Vital Capacity (FVC) result of the pulmonary function testing was to be used as a pulmonary function parameter. It was performed via standard office spirometry. It was calculated as an absolute value (in liters) and as a percentage (compared to the normal population data) It was to be used as a validation method to ensure patients did not have a former yet undiagnosed respiratory disease and to validate the presence of abnormal Peak Expiratory Flow (PEF) values.
Time Frame: Forced Vital Capacity was evaluated at the follow-up evaluation, which was performed 1 month post- baseline evaluation.
Population: Due to cooperation difficulties and/or differences above 10% in repeated testing, a total of 6 patients were excluded from the FVC evaluation.
Measure: Median (Full Range); unit: Percentage of Predicted Value
Arm/Group | Incentive Spirometer Group | Standard Care Group
Number analyzed (Participants) | 7 | 3
Percentage of Predicted Value | 80 [52 to 123] | 95 [58 to 103]

6. Secondary Outcome: Mortality
Description: Mortality will be accepted as a secondary outcome measure, in patients who may not survive until the monthly evaluation for any reason.
Time Frame: Mortality evaluation will include the time period of one month after hospital discharge. The total evaluation duration will also include the hospitalization period (which is considered an average of 7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Incentive Spirometer Group | Standard Care Group
Number analyzed (Participants) | 10 | 4
Participants | 0 | 0

7. Secondary Outcome: Discharge to Follow-up Duration (Days)
Description: The duration between the baseline evaluation at the time of hospital discharge and the first follow-up is defined as "Discharge to Follow-up Duration". There happens a time difference between post-one month evaluation and this definition, due to appointment dates; the exact one month time for a patient happening to be within weekend days or due to delays in respiratory testing. This could be observed by the time range of patients given here, as some (as seen in patients arriving within 13 days) had come to the hospital earlier, while some ( in the other end of the group, such as those arriving at 41st day) had either arrived late or could not be evaluated with respiratory function testing due to appointment or testing issues up to the day mentioned.
Time Frame: The time frame for "Discharge to Follow-up Duration" consisted of up to two months post-baseline evaluation. When a patient had arrived for the first follow-up evaluation, the time difference between baseline evaluation and this re-evaluation was noted.
Measure: Median (Full Range); unit: Days
Arm/Group | Incentive Spirometer Group | Standard Care Group
Number analyzed (Participants) | 10 | 4
Days | 31 [13 to 41] | 5 [3 to 13]

ADVERSE EVENTS:
Time Frame: The adverse event data were collected between the hospital admission time and the follow-up evaluation date. The follow-up evaluation was performed one month after hospital discharge and the median hospitalization duration was 8 days (3-18 full range). This accounts for a minimum of 33 days for the patient with the short follow-up and 48 days for the longest follow-up, regarding adverse data collection.
Arm/Group | Incentive Spirometer Group | Standard Care Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/4
Other Adverse Events (participants affected / at risk) | 0/10 | 0/4

LIMITATIONS AND CAVEATS:
All patients (n=84) admitted to the ward between these dates were evaluated for the study. Thirty-five patients were found suitable for the study. More than half of the suitable patients (n=21) refused to participate and thus were excluded from the study. This unexpected refusal to participation was the main limitation of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT04826731/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT04826731/ICF_001.pdf